CLINICAL TRIAL: NCT02286557
Title: Testing the Effects of Methylphenidate on Cognitive Fatigue in Multiple Sclerosis: a Double-blind, Placebo-controlled, Randomized Clinical Trial
Brief Title: Testing the Effects of Methylphenidate on Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Silvana Costa, Research Scientist, Kessler Foundation
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PP2280
Record Dates: First submitted 2014-10-16; First posted 2014-11-10 (Estimated); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Fatigue in Multiple Sclerosis
Keywords: Methylphenidate; Multiple Sclerosis; Cognitive Fatigue
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Arm 1 will undergo four weeks of treatment with MP extended-release (20 mg/day in the morning). Following the four weeks of treatment, all assessments performed at baseline will be repeated. To minimize practice effects, alternate versions of the neuropsychological tests will be used wherever available. A 7-day washout period will follow in which no medication will be administered. Following the washout period, Arm 1 will undergo four weeks of placebo. This will be followed by a final assessment consisting of measures of fatigue, cognitive functioning, and physical disability.
  Interventions: Drug: Methelphenidate; Drug: Placebo
- Arm II (Experimental): Arm 2 will undergo four weeks of placebo (in the morning). Following the four weeks of placebo, all assessments performed at baseline will be repeated. To minimize practice effects, alternate versions of the neuropsychological tests will be used wherever available. A 7-day washout period will follow in which no medication will be administered. Following the washout period, Arm 2 will undergo four weeks of treatment with MP extended-release (20mg/day). This will be followed by a final assessment consisting of measures of fatigue, sleep quality, cognitive functioning, and physical disability.
  Interventions: Drug: Methelphenidate; Drug: Placebo

INTERVENTIONS:
Drug: Methelphenidate — All participants will undergo 4 weeks of treatment with Methelphenidate and 4 weeks of placebo
Drug: Placebo

SUMMARY:
Up to 95% of individuals with Multiple Sclerosis report experiencing cognitive fatigue, characterized by a lack of energy, feelings of exhaustion, an the perception that one is unable to partake in daily activities. The goal of this project is to test whether methylphenidate (MP), a well-known psychostimulant, can effective treat fatigue experienced by individuals with MS.

The current study will test the effect of MP on MS fatigue through a clinical trial. Every participant in the study will be exposed to both the drug and the placebo for a period of time. Both the investigators and participants will be unaware whether participants are receiving the drug or the placebo.

Upon successful completion of the study, physicians will be able to evaluate the potential prescription of MP to treat fatigue in persons with MS based on solid research evidence. Importantly, MP is already an FDA approved widely used medication in multiple clinical populations.

DETAILED DESCRIPTION:
As highlighted by the National Clinical Advisory Board of the National Multiple Sclerosis Society (NMSS), "fatigue is the most common MS (multiple sclerosis) symptom", affecting up to 95% of individuals. Higher levels of cognitive fatigue have been associated with poorer quality of life (Amato & Portaccio, 2012) and increased disability (Lapierre & Hum, 2007), negatively affecting wellness. Several medications are currently prescribed to individuals with MS who suffer from fatigue, such as amantadine and modafinil. However, the effect of these medications on decreasing fatigue levels in individuals with MS is suboptimal (e.g. Stankoff et al., 2005). At the same time, there is overwhelming evidence showing that methylphenidate is effective at relieving fatigue in individuals with cancer (Minton et al., 2013), human immunodeficiency virus (Breitbart, Rosenfeld, Kaim, & Funesti-Esch, 2001), Parkinson's disease (Devos et al., 2013) and chronic fatigue syndrome (CFS) (Blockmans et al., 2006). For example, individuals with CFS reported decreased fatigue levels (as measured with a visual analogue scale) when taking MP (Blockmans et al., 2006). Although MP has been demonstrated to be an effective fatigue-relieving drug in multiple clinical populations discussed above, the effect of MP on MS-related fatigue has not been objectively tested.

MP is a psychostimulant that acts by inhibiting presynaptic dopamine transporters leading to suppression of dopamine reuptake (Prommer, 2012). That is, due to reuptake suppression, more dopamine remains in the synapses. MP primarily affects the striatum (which receives dopamine neuron projections from the substantia nigra pars compacta) and subsequently the prefrontal cortex (PFC), which receives dopaminergic projections from the striatum (Volkow et al., 2001).

To our knowledge, the only randomized clinical trial using MP in persons with MS assessed the effect of this medication on attention, reporting significant improvements in cognitive task performance (PASAT) in the MP treatment group (Harel, Appleboim, Lavie, & Achiron, 2009) as compared to a placebo control group. While an expert opinion paper sponsored by the NMSS recommends the use of MP to treat fatigue (Expert Opinion Paper, 2006), to our knowledge, no clinical trials have been conduced to objectively test the effect of MP administration on fatigue in individuals with MS and support this recommendation. The current study will fill this void in the literature. Aim 1: We propose to test the efficacy of MP on decreasing self-reported fatigue in individuals with MS in a double blind placebo controlled randomized clinical trial (DBRCT). Aim 2: We will also examine the effects of MP on cognitive functioning. Based on the existing literature on MP (Bales, Wagner, Kline, & Dixon, 2009; Harel et al., 2009), we expect that MP will enhance processing speed and attention, with little impact on other cognitive functions such as memory or executive control.

Significance: Our DBRCT will be the first to empirically assess the efficacy of MP as a treatment of MS-related fatigue. The application of the stringent RCT methodology will result in Class I evidence supporting or refuting the efficacy MP as a fatigue-relieving drug. The amelioration of fatigue in MS will have a significant positive impact on the MS population, given the prevalence and negative effects of fatigue.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Multiple Sclerosis
2. Age: 18-65 years old

Exclusion Criteria:

1. Participants must be free of: corticosteroids, cannot be currently taking modafinil, amantadine or other psychostimulants.
2. Participants must be MS relapse free at least during the previous 4 weeks.
3. Participants cannot consume more than ≧300mg of caffeine per day.
4. Thyroid disease
5. Anemia
6. Decreased vitamin D.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2014-10; Primary Completion 2025-02-28 (Actual); Study Completion 2025-03-04 (Actual)

PRIMARY OUTCOMES:
Fatigue - Modified Fatigue Impact Scale | baseline, day 30 and day 68
  Changes on fatigue levels from baseline, will be assess after 4 weeks, and after 10 weeks of the duration of the study.

SECONDARY OUTCOMES:
Processing Speed - Symbol Digit Modalities Test | baseline, day 30 and day 68
  Changes on Processing speed from baseline, will be assess after 4 weeks, and after 10 weeks of the duration of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, East Hanover, New Jersey, United States